CLINICAL TRIAL: NCT00671463
Title: Leak Elimination After Pancreatic Stenting, a Randomized Controlled Trial
Brief Title: Pancreatic Stent to Prevent Leak After Distal Pancreatectomy
Acronym: LEAPS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Anticipated high risk of pancreatitis
Sponsor: Massachusetts General Hospital (Other)
Collaborators: American Society for Gastrointestinal Endoscopy (Other)
Responsible Party: Principal Investigator, William R. Brugge, MD, Director of Gastrointestinal Endoscopy, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2007P000965
Record Dates: First submitted 2008-05-01; First posted 2008-05-05 (Estimated); Last update posted 2013-06-11 (Estimated); Status verified 2013-06

CONDITIONS: Pancreatic Surgery; Pancreatic Duct Stenting; Pancreatic Cancer; Distal Pancreatectomy; Pancreatic Diseases; Pancreatic Cyst; Pancreatic Ducts
Keywords: Pancreas surgery; Pancreatic adenocarcinoma; Pancreatic neuroendocrine tumor; Pancreatic duct stenting
MeSH Terms: conditions — Pancreatic Neoplasms; Pancreatic Diseases; Pancreatic Cyst; Adenoma, Islet Cell

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Pre-operative pancreatic duct stenting
  Interventions: Procedure: Pancreatic duct stenting
- 2 (No Intervention): Control group, no endoscopy and no stent pre-operatively

INTERVENTIONS:
Procedure: Pancreatic duct stenting — In the treatment arm, patients will have a pancreatic duct stent placed prior to having their distal pancreatectomy.
  Arms: 1

SUMMARY:
The purpose of this study is to investigate an intervention to prevent complications after pancreas surgery. The goal is to determine if placing a stent into the pancreatic duct before surgery will decrease or prevent leaking from the pancreatic duct after surgery. Leaks are common after pancreas surgery and can result in serious problems and post-operative pain. The study will compare two groups. One group will have the stent before surgery, and the other group will have standard pancreas surgery, no endoscopy, and no stent.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (greater than or equal to 18 years of age)
* Scheduled to undergo an elective laparoscopic or open distal pancreatectomy
* Willing to undergo pre-operative endoscopy
* Consenting to the procedure

Exclusion Criteria:

* Contraindication to abdominal surgery
* Contraindication to general anesthesia or distal pancreatectomy
* Contraindication to upper endoscopy or ERCP
* Prior history of gastric bypass or other abdominal surgery in whom the ampulla will not be accessible via routine ERCP
* Ongoing pancreatitis
* Pancreatic necrosis or abscess
* History of sphincter of Oddi dysfunction
* History of ERCP-induced pancreatitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-04; Primary Completion 2010-04 (Estimated)

PRIMARY OUTCOMES:
Pancreatic leak | Post-operative day 3

SECONDARY OUTCOMES:
Peritoneal fluid analysis | Daily
Serum biochemical analysis | Daily
Clinical outcomes | Daily

CONTACTS AND LOCATIONS:
Overall Officials: Field F Willingham, MD, MPH, Study Director — MGH; Denise W Gee, MD, Study Director — MGH; Sevdenur Cizginer, MD, Study Director — MGH; David W Rattner, MD, Principal Investigator — MGH; William R Brugge, MD, Principal Investigator — MGH
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States